CLINICAL TRIAL: NCT06186466
Title: Assessing Factors Influencing Violence Intent Among Families in Emergency Departments: A Multicenter Cross-Sectional Study
Brief Title: Family Violence Intent in Emergency Departments: A Multicenter Study
Status: Completed | Type: Observational
Sponsor: Kilis 7 Aralik University (Other)
Responsible Party: Principal Investigator, İslam Elagöz, Researcher Asisstan, Kilis 7 Aralik University
Other Study IDs: kilis7aralıkUn21
Record Dates: First submitted 2023-12-16; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Violence; Nurse-Patient Relations; Violence, Physical

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observational Survey and Analysis — This study does not involve a clinical or medical intervention. Instead, it employs an observational survey method to gather data from family members of patients who visited the Health Sciences University Van Training and Research Hospital's emergency department between December 1, 2023, and June 1, 2024. The study aims to use logistic regression analysis to identify factors influencing the intent of violence against healthcare professionals. The survey includes structured questionnaires and scales developed based on theoretical frameworks and previous research. The gathered data will be statistically analyzed using the G*Power software to assess the significance and impact of various factors on the propensity for violence.

SUMMARY:
This study addresses the growing issue of violence against healthcare professionals, particularly in emergency departments. It highlights the increasing prevalence of violence in healthcare settings worldwide, affecting over 50% of workers, with rates higher in developing countries. The text reviews factors contributing to violence, including poor communication, substandard care, and the stress experienced by patients' families. It notes that nearly 100% of emergency nurses face verbal or physical assaults. The research emphasizes the need to understand violence from the perspective of patients' families, a relatively unexplored area. By identifying the factors influencing their violent intentions, effective prevention measures can be developed, improving safety and working conditions for healthcare professionals.

DETAILED DESCRIPTION:
"Violence is a universal issue that harms the social fabric, threatening the lives, health, peace, and happiness of people in society. It negatively affects all communities and countries worldwide. Incidences of violence are increasingly visible in streets, schools, homes, and workplaces (WHO 2002). The International Labour Organization (ILO), International Council of Nurses (ICN), World Health Organization (WHO), and Public Services International (PSI) define workplace violence as 'the intentional use of physical force or power, threatened or actual, against oneself, another person, or against a group or community, that either results in or has a high likelihood of resulting in injury, death, psychological harm, maldevelopment, or deprivation' (Somani 2021). Over the last decade, there has been a noticeable increase in violence in healthcare settings (WMA 2020). Although underreported, it is estimated that over 50% of healthcare workers worldwide have experienced violence (Pompeii 2015), with this rate rising to 70% in developing countries (Belayachi 2010). Studies in Turkey support these findings (Polat 2019). A 2020 study in Turkey showed that 76% of doctors experienced violence at least once in their career (Çevik 2020). Another study in Turkey in 2020 indicated that 79% of healthcare workers experienced violence within the last year (Oğuz 2020). Research shows that emergency department healthcare workers are more frequently subjected to violence by patients and their family members (Kowalenko 2013; Şanlıtürk 2021). One study reported that 100% of emergency nurses experienced verbal assault, and 82.1% experienced physical assault within a year (May 2002). A Turkish study showed that about 75% of emergency department healthcare workers had been exposed to violence (Kaya 2016). Violence in emergency departments is influenced by various factors related to administration, staff, security, environment, patients, or their family members. For instance, lack of communication among healthcare professionals, poor quality of care, increased anxiety levels of patients' families, and stress due to a patient's critical condition can be contributing factors (AbuAlRub 2014).

Family members accompanying patients to emergency departments often exhibit violent tendencies due to increased stress and the aforementioned factors, leading to negative consequences. This violence results in injuries, additional work stress for healthcare workers, and reduced work efficiency, thereby lowering the quality of healthcare provided (Kowalenko 2013; Polat 2019). It also diminishes job satisfaction among healthcare workers and can lead to burnout (Polat 2019; Şanlıtürk 2021). Literature review shows that violence against healthcare workers has been well examined. Studies have demonstrated the frequency of violence healthcare professionals face, which professional groups are more often subjected to violence, and how characteristics such as educational level, gender, and professional experience of healthcare professionals affect their exposure to violence. The impact of security personnel, management, and institutional policies on violence in healthcare has also been explored (AbuAlRub 2014; Baykan 2015; da Silva 2015; Kitaneh 2012; Hanh 2013; Polat 2019; Kowalenko 2013; Pompeii 2015; Çevik 2020). However, research focusing on the perspectives of patients' families on violence in healthcare and factors influencing their violent tendencies and intentions towards healthcare staff is limited. This gap limits the effectiveness of measures to prevent violence against healthcare professionals and hinders the desired level of violence prevention in healthcare. Identifying the violent intentions of patients' families and the factors influencing them will contribute to the effectiveness of measures taken to prevent violence against healthcare professionals. This study aims to identify the intentions and influencing factors of violence by family members of patients presenting to emergency departments towards healthcare staff.

ELIGIBILITY:
Inclusion Criteria:

* Must be over 18 years old, Able to speak and write in Turkish, Without hearing or communication impairments, Without mental disabilities, Family members related by blood or marriage to patients presenting to the emergency department of the hospital where the study is conducted, Voluntarily willing to participate in the study.

Exclusion Criteria:

* Family members of patients whose condition becomes critical and are taken to the resuscitation room, Data from family members who decide to withdraw from the study at any stage after being included will not be considered in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population comprises family members of patients admitted to the emergency department of the hospital where the research is conducted. Participants are adults over 18 years old who are fluent in Turkish and do not have any hearing, communication, or mental disabilities. The population includes those who are either blood relatives or related by marriage to the patients. All participants are included based on their voluntary consent to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Part 1: Demographic Information Form | up to 9 weeks
  The first part of the data collection form includes questions aimed at determining the age, gender, educational status, marital status, family type, and occupation of the family members. This section also contains questions to ascertain any history of violence in the patient's social life and whether they have received psychological treatment for violence.
Intent to Commit Violence Against Healthcare Workers Scale | up to 9 weeks
  Developed by Şanlıtürk and Boy based on Ajzen's Theory of Planned Behavior, this 15-item Likert scale assesses the intent to commit violence and its influencing factors: past experiences, attitude towards behavior, subjective norms, and perceived behavioral control. The scale uses a 5-point scoring system, with reverse scoring for specific items.
Part 3: Factors Influencing Intent to Commit Violence Against Healthcare Professionals Form | up to 9 weeks
  Created after reviewing various sources, this form contains 22 structured questions on a 5-point Likert scale to identify factors influencing family members' intent to commit violence against healthcare professionals. The form's content validity was assessed by healthcare experts, resulting in a Content Validity Index (CVI) of 0.96, indicating suitability for this research.

CONTACTS AND LOCATIONS:
Overall Officials: islam elagöz, Study Chair — kils 7 aralık University
Locations (1):
- Islam Elagöz, Kilis, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We do not plan to make individual participant data (IPD) available to other researchers. This decision is based on concerns regarding the privacy and confidentiality of the study participants. The sensitive nature of the data collected in this study, especially considering it involves family members of patients in emergency departments, necessitates strict adherence to privacy standards. Therefore, to ensure the protection of our participants' privacy and to comply with ethical standards, IPD will not be shared or made accessible for external use.